CLINICAL TRIAL: NCT01950481
Title: A Phase I, Open Label, Multi-center, Single Dose Study to Evaluate the Pharmacokinetics of LDK378 in Subjects With Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: Effect of Hepatic Impairment on LDK378 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2110
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-12

CONDITIONS: Normal Hepatic Function; Impaired Hepatic Function
Keywords: LDK378; pharmacokinetics; hepatic impairment
MeSH Terms: interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal Hepatic Function (Experimental): Subjects with normal hepatic function
  Interventions: Drug: LDK378
- Mild Hepatic Impairment (Experimental): Subjects with mild hepatic impairment
  Interventions: Drug: LDK378
- Moderate Hepatic Impairment (Experimental): Subjects with moderate hepatic impairment
  Interventions: Drug: LDK378
- Severe Hepatic Impairment (Experimental): Subjects with severe hepatic impairment
  Interventions: Drug: LDK378

INTERVENTIONS:
Drug: LDK378 — Oral LDK378 750 mg once

SUMMARY:
Pharmacokinetics and safety of 750 mg of LDK378 given once orally in subjects with impaired hepatic function and healthy subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria (all groups):

* Male Subjects between 18-70 years of age
* Female subjects between 18-70 years of age who are postmenopausal or sterile
* Body Mass Index (BMI) of 18.0- 36.0 kg/m2, with body weight ≥ 50 kg.

Inclusion (group mild, moderate and severe hepatic impairment):

- Subjects with confirmed cirrhosis

Exclusion Criteria (all groups):

* impaired cardiac function
* concurrent severe and/or uncontrolled medical conditions

Exclusion Criteria (moderate, mild and severe groups):

* Clinical evidence of severe ascites
* Use of PPIs within 10 days prior to 2 days after LDK378 dosing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
LDK378 pharmacokinetic parameters (Tmax) | 18 Days
  Evaluate the pharmacokinetics of a single dose of LDK378 in subjects with impaired hepatic function as compared to healthy subjects
LDK378 pharmacokinetic parameters ( Cmax) | 18 Days
  Evaluate the pharmacokinetics of a single dose of LDK378 in subjects with impaired hepatic function as compared to healthy subjects
LDK378 pharmacokinetic parameters ( AUClast) | 18 Days
  Evaluate the pharmacokinetics of a single dose of LDK378 in subjects with impaired hepatic function as compared to healthy subjects
LDK378 pharmacokinetic parameters (AUCinf) | 18 Days
  Evaluate the pharmacokinetics of a single dose of LDK378 in subjects with impaired hepatic function as compared to healthy subjects
LDK378 pharmacokinetic parameters (T1/2) | 18 Days
  Evaluate the pharmacokinetics of a single dose of LDK378 in subjects with impaired hepatic function as compared to healthy subjects
LDK378 pharmacokinetic parameters (CL/F) | 18 Days
  Evaluate the pharmacokinetics of a single dose of LDK378 in subjects with impaired hepatic function as compared to healthy subjects
LDK378 pharmacokinetic parameters (Vz/F) | 18 Days
  Evaluate the pharmacokinetics of a single dose of LDK378 in subjects with impaired hepatic function as compared to healthy subjects

SECONDARY OUTCOMES:
Number of subjects with Adverse events | after informed consent is signed, 30 days after last dose
  Safety will be determined by the frequency of adverse events and the frequency of laboratory toxicities.
Plasma protein binding of LDK378 | Day 1 predose, Day 1 6 hours postdose
  Plasma protein binding of LDK378

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - DaVita Clinical Research-Denver, Lakewood, Colorado
  - Avail. Clinical Research, LLC, DeLand, Florida
  - Clinical Research of Miami, INC CLDK378A2110, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota

REFERENCES:
- See also: Results for CLDK378A2110 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16555